CLINICAL TRIAL: NCT05840289
Title: FRILLY: A Retrospective Single-centre Study on Fractionated Rituximab to Avoid Lysis Syndrome in Aggressive B-Lymphoma
Brief Title: A Study on Fractionated Rituximab to Avoid Lysis Syndrome in Aggressive B-Lymphoma
Acronym: FRILLY
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Noémie Lang, Principal Investigator, University Hospital, Geneva
Other Study IDs: 2020-01659
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Aggressive B-Cell Non-Hodgkin Lymphoma
Keywords: Aggressive B-cell non-Hodgkin lymphoma; tumor lysis syndrome; fractionated rituximab; prevention
MeSH Terms: conditions — Tumor Lysis Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: fractionated first dose rituximab — Patients at high-risk to develop tumor lysis syndrome received a initial fractionated dose of rituximab over 2 or 3 days

SUMMARY:
Tumour lysis syndrome (TLS) occurs as a consequence of the rapid destruction of malignant cells, spontaneously and/or in response to cytotoxic agents and immunotherapies. TLS is a feature of highly proliferative diseases with heavy tumor burden, such as high-grade non-Hodgkin lymphomas (NHL, typically Burkitt's lymphoma). We evaluated fractionating first rituximab dose to prevent TLS in a real-life B-cell NHL cohort of patients treated at University Hospital of Geneva between 2010 and 2020.

DETAILED DESCRIPTION:
Tumour lysis syndrome (TLS) occurs as a consequence of the rapid destruction of malignant cells, spontaneously and/or in response to cytotoxic agents and immunotherapies. TLS is a feature of highly proliferative diseases with heavy tumor burden, such as acute lymphoblastic leukemia (B-ALL) and high-grade non-Hodgkin lymphomas (NHL, typically Burkitt's lymphoma). TLS usually develop during the first week of treatment due to the sudden release of intracellular ions, nucleic acids and protein metabolites. These metabolic disturbances can manifest as hyperuricemia, hyperkaliemia, hyperphosphatemia, hypocalcemia and uremia, exposing the patient to acute renal insufficiency, lactic acidosis and ultimately death in the absence of appropriate management.

In order to make them more practical and reproducible, TLS criteria were modified in 2004 by Cairo and Bishop, who also developed a grading classification as: 1) biochemical TLS occurring 3 days before to 7 days after the start of therapy, and 2) clinical TLS in case of seizure, cardiac arrhythmia or significant acute renal injury (AKI). TLS is burdened with significant morbidity and mortality.

Historically, TLS incidence among high-grade non-Hodgkin's lymphoma (NHL) patients was reported in as high as 42% of cases, with 6% of clinically significant TLS. In a more recent multicentric retrospective analysis performed on 722 patients (37% NHL, 36% ALL, 27% AML), 5.2 % of the patients developed TLS, and among them 25% required intensive care unit admission with a relative mortality rate of 15%.

Rituximab (Mabthera®, Swissmedic 54378) is a therapeutic monoclonal antibody that binds with high affinity to cells expressing the CD20 antigen found on the surface of malignant and normal B cells, inducing complement-dependent and antibody-dependent cellular cytotoxicity. Approved in 1997 for the treatment of CD20-positive B-cell low-grade NHL, rituximab is now widely used in all the spectrum of B-cell malignancies. Initially administered on a weekly schedule for a total of 4 to 8 infusions, rituximab is currently infused together with other cytotoxic agents every 3 to 4 weeks. Rituximab may cause a massive cytolysis of B-cells in some patients leading to an acute onset TLS. Notably, TLS was reported as the second significant safety signal after rituximab administration in 1998.

Since the development of uricolytic agents (rasburicase), TLS incidence has significantly been reduced. Nevertheless, early risk-stratification and initiation of a comprehensive supportive care are mandatory in TLS. The mainstays of TLS prophylaxis and treatment include hydration and diuresis, control of hyperuricaemia with xanthine oxidase inhibitors blocking endogenous uric acid production from purine nucleotides (eg. allopurinol) or uricolytic agents (rasburicase), and vigilant monitoring of electrolyte abnormalities.

In addition, preemptive strategies of tumor debulking were developed such as steroids or low-dose chemotherapy prophase or gradual dose ramp-up of the cytotoxic agent as exemplified with the administration of the Bcl2 inhibitor Venetoclax in chronic lymphocytic leukemia.

To prevent TLS, but also other side effects such as allergy and cytokine-release syndrome during the first administration of rituximab, a few studies suggested the use of a fractionated and dose ramp-up schedule of rituximab administration in B-cell malignancies. In Geneva University Hospital (HUG), this strategy was widely applied to most cases of patients having a B-cell malignancy at high-risk for TLS since the publication of these pioneer studies. We aim at investigating the incidence and severity of TLS in high-grade B-cell lymphoma patients treated at HUG over the last ten years.

Main objective To evaluate the incidence of biochemical lysis syndrome (LTLS) and clinical lysis syndrome (CTLS) in patients receiving fractionated Rituximab infusion for high-grade B-cell lymphoma.

Inclusion

• Newly diagnosed or relapsing histologically proven B-cell lymphoma patients treated with fractionated Rituximab infusion, considered as ≥ 2 consecutive infusions, at least 24 hours apart

Exclusion

* Unproven histologically B-cell lymphoma
* Patients who receive a single day Rituximab infusion
* Patients under long-term dialysis before Rituximab started
* Age ≤ 18 years
* Absence of written informed consent

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or relapsing histologically proven high-grade B-cell lymphoma patients treated with fractionated Rituximab infusion, considered as ≥ 2 consecutive infusions, at least 24 hours apart

Exclusion Criteria:

* Unproven histologically high-grade B-cell lymphoma
* Patients who receive a single day Rituximab infusion
* Patients under long-term dialysis before Rituximab started
* Age ≤ 18 years
* Absence of written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: histologically proven high-grade B-cell lymphoma patients
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of clinical lysis syndrome (CTLS) in patients receiving fractionated Rituximab infusion for high-grade B-cell lymphoma. | 10 days (day -2 and day + 7 after first rituximab infusion)
  To evaluate the incidence of clinical tumor lysis syndrome (CTLS) in patients receiving fractionated Rituximab infusion for high-grade B-cell lymphoma.

SECONDARY OUTCOMES:
Incidence of biochemical lysis syndrome (LTLS) in patients receiving fractionated Rituximab infusion for high-grade B-cell lymphoma. | 10 days (day -2 and day + 7 after first rituximab infusion)
  To evaluate the incidence of biochemical tumor lysis syndrome (LTLS) in patients receiving fractionated Rituximab infusion for high-grade B-cell lymphoma.

CONTACTS AND LOCATIONS:
Overall Officials: Noemie Lang, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospital Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All anonymised IPD that underlie results in a publication will be shared upon request with other researchers.
  Types of supporting information that will be shared, in addition to the individual participant data set and data dictionaries will include the study protocol, informed consent form and clinical study report
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 10 years
Access Criteria: Upon reasonable scientific request